CLINICAL TRIAL: NCT02910583
Title: Phase 2 Study of the Combination of Ibrutinib Plus Venetoclax in Subjects With Treatment-naïve Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Ibrutinib Plus Venetoclax in Subjects With Treatment-naive Chronic Lymphocytic Leukemia /Small Lymphocytic Lymphoma (CLL/SLL)
Acronym: Captivate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCYC-1142-CA; 2016-002293-12 (EudraCT Number)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Leukemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants with confirmed undetectable minimal residual disease (uMRD) in the MRD cohort are triple masked.
  Allocation was not randomized for the Fixed Duration (FD) cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Fixed Duration (FD) Cohort: Open Label Ibrutinib + Venetoclax (Experimental): Participants receive 420 mg of single-agent ibrutinib for first 3 cycles followed by ibrutinib plus venetoclax combination treatment (ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule) for 12 cycles (a cycle is defined by 28 days) or until disease progression or unacceptable toxicity.
  Interventions: Drug: ibrutinib; Drug: venetoclax
- MRD Cohort/Confirmed Undetectable MRD (uMRD): Randomized to Ibrutinib (Blinded) (Experimental): Participants receive 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase).
  Participants with confirmed uMRD are randomized to receive ibrutinib 420 mg orally once daily on a continuous schedule until MRD-positive relapse, disease progression (PD), or unacceptable toxicity.
  After MRD-positive relapse or disease progression (PD) by iwCLL criteria, participants can reintroduce 400 mg venetoclax with a 5-week ramp up. If venetoclax is to be reintroduced, venetoclax treatment is to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) until PD or unacceptable toxicity.
  Interventions: Drug: ibrutinib; Drug: venetoclax
- MRD Cohort/Confirmed uMRD: Randomized Placebo (Blinded) (Placebo Comparator): Participants receive 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase).
  Participants with confirmed uMRD are randomized to receive placebo orally once daily on a continuous schedule until MRD-positive relapse, PD or unacceptable toxicity.
  If MRD-positive relapse or PD is confirmed after restaging per iwCLL criteria, participants can first reintroduce oral daily ibrutinib with the option of subsequently reintroducing 400 mg venetoclax with a 5-week ramp up, if subsequent disease relapse per iwCLL criteria occurs after ibrutinib reintroduction. If venetoclax is to be reintroduced, venetoclax treatment is to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) until PD or unacceptable toxicity.
  Interventions: Drug: ibrutinib; Drug: venetoclax; Drug: Placebo
- MRD Cohort/uMRD Not Confirmed: Randomized to Ibrutinib (Open-Label) (Experimental): Participants receive 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre randomization phase).
  Participants with uMRD not confirmed are randomized to receive open-label ibrutinib 420 mg orally once daily on a continuous schedule until PD or unacceptable toxicity.
  In case of confirmed PD after restaging per iwCLL criteria, participants can continue ibrutinib and reintroduce venetoclax treatment. If venetoclax is to be reintroduced, venetoclax treatment is to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) until PD or unacceptable toxicity.
  Interventions: Drug: ibrutinib; Drug: venetoclax
- MRD Cohort/uMRD Not Confirmed: Randomized Ibrutinib + Venetoclax (Open-Label) (Experimental): Participants receive 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre randomization phase).
  Participants with uMRD not confirmed are randomized to receive open-label ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity. Venetoclax was allowed for administration up to 2 years cumulatively from first dose started in the pre-randomization phase to last dose in the randomization phase.
  Interventions: Drug: ibrutinib; Drug: venetoclax

INTERVENTIONS:
Drug: ibrutinib — ibrutinib administered orally once daily (three 140 mg capsules)
Drug: venetoclax — venetoclax tablets will be administered orally once daily starting with a 5 week ramp up of 20 mg, 50 mg, 100 mg, 200 mg and 400 mg. After ramp up, venetoclax will be administered at 400 mg.
Drug: Placebo — placebo capsules to match ibrutinib administered orally once daily
  Arms: MRD Cohort/Confirmed uMRD: Randomized Placebo (Blinded)

SUMMARY:
This is a multicenter, 2-cohort Phase 2 study assessing both minimal residual disease (MRD)-guided discontinuation and fixed duration therapy with the combination of ibrutinib + venetoclax in subjects with treatment-naïve CLL or SLL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL/SLL that meets 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) diagnostic criteria (Hallek et al), with active disease meeting at least 1 IWCLL criteria for requiring treatment.
* Measurable nodal disease by computed tomography (CT)
* Adequate hepatic, and renal function
* Adequate hematologic function
* absolute neutrophil count >750/µL
* platelet count >30,000 /μL
* hemoglobin >8.0 g/dL

Exclusion Criteria:

* Any prior therapy used for treatment of CLL/SLL
* Known allergy to xanthine oxidase inhibitors and/or rasburicase for subjects at risk for tumor lysis syndrome (TLS)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (46):
- United States (14):
  - City of Hope /ID# 1142-0047, Duarte, California
  - Moores Cancer Center at UC San Diego /ID# 1142-0241, La Jolla, California
  - UC Irvine Medical Center - Chao Family Comprehensive Cancer Center /ID# 1142-0008, Orange, California
  - Norton Cancer Center /ID# 1142-0071, Louisville, Kentucky
  - Rutgers Cancer Institute of New Jersey /ID# 1142-1193, New Brunswick, New Jersey
  - Northwell Health/Long Island Jewish Hospital /ID# 1142-0350, New Hyde Park, New York
  - New York Presbyterian Hospital/Weill Cornell Med College /ID# 1142-0200, New York, New York
  - University of Rochester Cancer Center /ID# 1142-0127, Rochester, New York
  - Charlotte-Mecklenberg Hospital, Carolinas Healthcare System, Levine Cancer Inst /ID# 1142-0733, Charlotte, North Carolina
  - Cleveland Clinic Foundation /ID# 1142-0739, Cleveland, Ohio
  - University of Pennsylvania /ID# 1142-0069, Philadelphia, Pennsylvania
  - Tennessee Oncology - Chattanooga /ID# 1142-0123, Chattanooga, Tennessee
  - MD Anderson Cancer Center /ID# 1142-0032, Houston, Texas
  - Swedish Cancer Institute /ID# 1142-0114, Seattle, Washington
- Australia (7):
  - St George Hospital /ID# 1142-0654, Kogarah, New South Wales
  - Flinders Medical Centre /ID# 1142-0163, Bedford Park, South Australia
  - Monash Medical Centre /ID# 1142-0556, Clayton, Victoria
  - Peter MacCallum Cancer Centre-East Melbourne /ID# 1142-0633, East Melbourne, Victoria
  - St Vincent's Hospital Melbourne /ID# 1142-0501, Fitzroy, Victoria
  - Frankston Hospital /ID# 1142-0715, Frankston, Victoria
  - Austin Health /ID# 1142-0170, Heidelberg, Victoria
- Italy (7):
  - Ospedale San Raffaele IRCCS /ID# 1142-0523, Milan, Lombardy
  - Ospedale Policlinico San Martino /ID# 1142-0903, Genova
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 1142-0581, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 1142-0524, Modena
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 1142-0582, Novara
  - Azienda Ospedaliera di Padova /ID# 1142-1175, Padua
  - Azienda USL di Piacenza - Ospedale Guglielmo da Saliceto /ID# 1142-1182, Piacenza
- New Zealand (4):
  - Middlemore Hospital /ID# 1142-0662, Otahuhu, Auckland
  - Christchurch Hospital /ID# 1142-0589, Christchurch, Canterbury
  - Palmerston North Hospital /ID# 1142-0585, Palmerston North, Manawatu-Wanganui
  - North Shore Hospital /ID# 1142-0663, Auckland
- Poland (5):
  - Malopolskie Centrum Medyczne /ID# 1142-0364, Krakow, Lesser Poland Voivodeship
  - Duplicate_Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie /ID# 1142-0590, Lublin, Lublin Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. ks. B. /ID# 1142-0592, Brzozów, Podkarpackie Voivodeship
  - Samodzielny Publiczny Szpital Klinczny Nr-1- Akademickie Cenrum Klinic /ID# 1142-0529, Gdansk, Pomeranian Voivodeship
  - Medical Univ. of Lodz and Copernicus Memorial Hospital /ID# 1142-0531, Lodz
- Spain (9):
  - Hospital Duran i Reynals /ID# 1142-0604, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda /ID# 1142-0536, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra /ID# 1142-1197, Pamplona, Navarre
  - Hospital Clinic de Barcelona /ID# 1142-0533, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 1142-0535, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 1142-1196, Granada
  - Hospital Universitario Ramon y Cajal /ID# 1142-0874, Madrid
  - Hospital Universitario 12 de Octubre /ID# 1142-0864, Madrid
  - Hospital Clinico Universitario de Salamanca /ID# 1142-0790, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
Supporting Information: Study Protocol, SAP, CSR
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Moreno C, Solman IG, Tam CS, Grigg A, Scarfo L, Kipps TJ, Srinivasan S, Mali RS, Zhou C, Dean JP, Szafer-Glusman E, Choi M. Immune restoration with ibrutinib plus venetoclax in first-line chronic lymphocytic leukemia: the phase 2 CAPTIVATE study. Blood Adv. 2023 Sep 26;7(18):5294-5303. doi: 10.1182/bloodadvances.2023010236. PMID 37315225
- [Derived] Wierda WG, Allan JN, Siddiqi T, Kipps TJ, Opat S, Tedeschi A, Badoux XC, Kuss BJ, Jackson S, Moreno C, Jacobs R, Pagel JM, Flinn I, Pak Y, Zhou C, Szafer-Glusman E, Ninomoto J, Dean JP, James DF, Ghia P, Tam CS. Ibrutinib Plus Venetoclax for First-Line Treatment of Chronic Lymphocytic Leukemia: Primary Analysis Results From the Minimal Residual Disease Cohort of the Randomized Phase II CAPTIVATE Study. J Clin Oncol. 2021 Dec 1;39(34):3853-3865. doi: 10.1200/JCO.21.00807. Epub 2021 Oct 7. PMID 34618601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 39 centers in the United States (US), Australia, New Zealand, Spain, and Italy.
Pre-assignment Details: Upon completion of a pre-randomization phase, participants in the MRD Cohort with confirmed undetectable minimal residual disease (uMRD) were randomized to blinded ibrutinib or placebo. Participants in the MRD Cohort with uMRD not confirmed were randomized to open-label ibrutinib or open-label ibrutinib + venetoclax.
Groups:
- Fixed Duration (FD) Cohort: All Treated: Participants received 420 mg of single agent ibrutinib for first 3 cycles followed by ibrutinib plus venetoclax combination treatment (ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule) for 12 cycles (a cycle is defined by 28 days) or until disease progression or unacceptable toxicity, whichever was earlier.
  Participants with confirmed progression per 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria after completion of the fixed duration regimen could be retreated with continuous single agent ibrutinib until disease progression or unacceptable toxicity, whichever was earlier, because it is an established standard of care for treatment of relapsed chronic lymphocytic leukemia (CLL).
  For participants who experienced durable efficacy after ibrutinib plus venetoclax (ie, time to progression after fixed duration regimen is completed of >2 years), the ibrutinib plus venetoclax fixed duration treatment regimen may have been repeated based on Investigator's clinical discretion and Medical Monitor's approval. Retreatment was for 15 cycles, until disease progression (PD) or unacceptable toxicity, whichever was earlier.
- Minimal Residual Disease (MRD) Cohort: All Treated: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants who completed the planned pre-randomization treatment were eligible to be randomized according to their confirmed undetectable minimal residual disease (uMRD) status: Participants with confirmed uMRD were randomized to receive blinded ibrutinib 420 mg or placebo orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg or open-label ibrutinib 420 mg plus venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. The venetoclax could be administered cumulative from pre-randomization to randomization phase at the dose of 400 mg/day for up to approximately 2 years, or earlier PD or unacceptable toxicity.
Period: Overall Study
Arm/Group | Fixed Duration (FD) Cohort: All Treated | Minimal Residual Disease (MRD) Cohort: All Treated
Started | 159 | 164
MRD Cohort/ Not Randomized | 0 (Not applicable to this cohort.) | 15
MRD Cohort/ Confirmed uMRD: Randomized to Ibrutinib (Blinded) | 0 (Not applicable to this cohort.) | 43
MRD Cohort/ Confirmed uMRD: Randomized Placebo (Blinded) | 0 (Not applicable to this cohort.) | 43
MRD Cohort/uMRD Not Confirmed: Randomized to Ibrutinib (Open-Label) | 0 (Not applicable to this cohort.) | 31
MRD Cohort/uMRD Not Confirmed: Randomized Ibrutinib + Venetoclax (Open-Label) | 0 (Not applicable to this cohort.) | 32
Completed (Participants who were on study when the sponsor closed the treatment arm or terminated the study and provided option to rollover to long term follow-up study.) | 133 | 150
Not Completed | 26 | 14
Not completed — Death | 7 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Other, Not Specified | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- FD Cohort: All Treated: Participants received 420 mg of single agent ibrutinib for first 3 cycles followed by ibrutinib plus venetoclax combination treatment (ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule) for 12 cycles (a cycle is defined by 28 days) or until disease progression or unacceptable toxicity, whichever was earlier.
  Participants with confirmed progression per 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria after completion of the fixed duration regimen could be retreated with continuous single agent ibrutinib until disease progression or unacceptable toxicity, whichever was earlier, because it is an established standard of care for treatment of relapsed chronic lymphocytic leukemia (CLL).
  For participants who experienced durable efficacy after ibrutinib plus venetoclax (ie, time to progression after fixed duration regimen is completed of >2 years), the ibrutinib plus venetoclax fixed duration treatment regimen may have been repeated based on Investigator's clinical discretion and Medical Monitor's approval. Retreatment was for 15 cycles, until disease progression (PD) or unacceptable toxicity.
- MRD Cohort: All Treated: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants who completed the planned pre-randomization treatment were eligible to be randomized according to their confirmed undetectable minimal residual disease (uMRD) status: Participants with confirmed uMRD were randomized to receive blinded ibrutinib 420 mg or placebo orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg or open-label ibrutinib 420 mg plus venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. The venetoclax could be administered cumulative from pre-randomization to randomization phase at the dose of 400 mg/day for up to approximately 2 years, or earlier PD or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | FD Cohort: All Treated | MRD Cohort: All Treated | Total
Number analyzed (Participants) | 159 | 164 | 323
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 114 | 123 | 237
  >= 65 years | 45 | 41 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 61 | 114
  Male | 106 | 103 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 16
  Not Hispanic or Latino | 149 | 150 | 299
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 147 | 147 | 294
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: MRD Cohort: 1-Year Disease-Free Survival (DFS) Rate in Confirmed uMRD Randomized Participants
Description: DFS is defined as time from randomization date to MRD-positive relapse, or disease progression per investigator assessment (per 2008 International Workshop for Chronic Lymphocytic Leukemia [IWCLL] criteria [Halleck et al]) or death from any cause, whichever occurred first. 1-year DFS estimated using Kaplan-Meier method at 12 months landmark time.
Time Frame: 1 year after randomization
Population: Confirmed uMRD Randomized Population: all participants who achieved confirmed MRD-negative clinical response at the end of the pre-randomization phase, randomized to either blinded placebo arm or blinded ibrutinib arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded): Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with confirmed uMRD were randomized to receive ibrutinib 420 mg orally once daily on a continuous schedule until MRD-positive relapse, PD, or unacceptable toxicity, whichever was earlier. After MRD-positive relapse or disease progression (PD) by iwCLL criteria, subjects can reintroduce 400 mg venetoclax with a 5-week ramp up. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative), or earlier PD or unacceptable toxicity.
- MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded): Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with confirmed uMRD were randomized to receive placebo orally once daily on a continuous schedule until MRD-positive relapse, PD or unacceptable toxicity, whichever was earlier. If MRD-positive relapse or PD is confirmed after restaging per iwCLL criteria, participants could first reintroduce oral daily ibrutinib with the option of subsequently reintroducing 400 mg venetoclax with a 5-week ramp up, if subsequent disease relapse per iwCLL criteria occurs after ibrutinib reintroduction. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative), or earlier PD or unacceptable toxicity.
Arm/Group | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded)
Number analyzed (Participants) | 43 | 43
percentage of participants | 100.0 [100.0 to 100.0] | 95.3 [82.7 to 98.8]
Statistical Analysis 1: Comparison: MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) vs MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded); Test type: Superiority; p = 0.1475, Z test — P-value is from Z test for the difference of two proportions based on Kaplan-Meier estimates with standard error of each arm computed using Greenwood's formula; Difference in Rates = 4.7, 95% CI 2-sided [-1.6 to 10.9] — comparison: ibrutininb vs. placebo

2. Primary Outcome: FD Cohort: Complete Response Rate (CRR; Complete Response/Complete Response With Incomplete Blood Count Recovery [CR/CRi]) Rate
Description: CR/CRi rate is defined as the percentage of participants achieving a best overall response of complete response (CR), CR with incomplete blood count recovery (CRi) per 2008 IWCLL criteria (halleck et al.) on or prior to initiation of subsequent antineoplastic therapy or, if applicable, reintroduction of study treatment, whichever occurred earlier.
Time Frame: From the first dose of ibrutinib to the first confirmed PD, for a median follow-up of 69.0 months.
Population: Per protocol, the primary analysis of the primary endpoint for the FD cohort was based on the FD Cohort, Non-Del 17p Population only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FD Cohort, Non-Del 17p Population: Participants in the FD cohort without del 17p abnormality (according to non-missing baseline fluorescent in situ hybridization [FISH] results) received 420 mg of single agent ibrutinib for first 3 cycles followed by ibrutinib plus venetoclax combination treatment (ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule) for 12 cycles (a cycle is defined by 28 days) or until PD or unacceptable toxicity, whichever was earlier.
- Fixed Duration (FD) Cohort: All Treated: Participants received 420 mg of single agent ibrutinib for first 3 cycles followed by ibrutinib plus venetoclax combination treatment (ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule) for 12 cycles (a cycle is defined by 28 days) or until disease progression or unacceptable toxicity, whichever was earlier.
  Participants with confirmed progression per 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria after completion of the fixed duration regimen could be retreated with continuous single agent ibrutinib until disease progression or unacceptable toxicity, whichever was earlier, because it is an established standard of care for treatment of relapsed chronic lymphocytic leukemia (CLL).
  For participants who experienced durable efficacy after ibrutinib plus venetoclax (ie, time to progression after fixed duration regimen is completed of >2 years), the ibrutinib plus venetoclax fixed duration treatment regimen may have been repeated based on Investigator's clinical discretion and Medical Monitor's approval. Retreatment was for 15 cycles, until disease progression (PD) or unacceptable toxicity.
Arm/Group | FD Cohort, Non-Del 17p Population | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 136 | 159
percentage of participants | 58.1 [49.8 to 66.4] | 57.2 [49.5 to 64.9]
Statistical Analysis 1: Comparison: FD Cohort, Non-Del 17p Population; Test type: Superiority; p < 0.0001, asymptotic test for binomial proportion — One-sided P-value from asymptotic test for the binomial proportion (CRR <= 37% vs CRR > 37%)

3. Secondary Outcome: MRD Cohort: CRR (CR/CRi Rate)
Description: CR/CRi rate is defined as the percentage of participants achieving a best overall response of CR or CRi per 2008 IWCLL criteria (Halleck et al.) on or prior to initiation of subsequent antineoplastic therapy or, if applicable, reintroduction of study treatment, whichever occurred earlier.
  Median follow up duration for the individual MRD Cohort treatment arms: Confirmed uMRD Ibrutinib arm 69.1 months; Confirmed uMRD Placebo arm 67.4 months; uMRD Not Confirmed Ibrutinib arm 47.9 months; uMRD Not Confirmed Ibrutinib + Venetoclax arm 47.9 months.
Time Frame: From the first dose of ibrutinib to the first confirmed PD, for an overall median follow-up of 67.0 months. (Median follow up duration for the individual MRD Cohort treatment arms listed above.)
Population: MRD Cohort - All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded): Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with confirmed uMRD were randomized to receive ibrutinib 420 mg orally once daily on a continuous schedule until MRD-positive relapse, PD, or unacceptable toxicity, whichever was earlier. After MRD-positive relapse or disease progression (PD) by iwCLL criteria, participants could reintroduce 400 mg venetoclax with a 5-week ramp up. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative), or earlier PD or unacceptable toxicity.
- MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. In case of confirmed PD after restaging per iwCLL criteria, participants could continue ibrutinib and reintroduce venetoclax treatment. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) or earlier PD or unacceptable toxicity.
- MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. In case of confirmed PD after restaging per iwCLL criteria, participants could continue ibrutinib and reintroduce venetoclax treatment. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) or earlier PD or unacceptable toxicity.
Arm/Group | MRD Cohort: All Treated | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded) | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 164 | 43 | 43 | 31 | 32
percentage of participants | 66.5 [59.2 to 73.7] | 79.1 [66.9 to 91.2] | 65.1 [50.9 to 79.4] | 77.4 [62.7 to 92.1] | 56.3 [39.1 to 73.4]

4. Secondary Outcome: MRD Cohort: Overall Response Rate (ORR)
Description: ORR, defined as the percentage of participants achieving a best overall response of protocol-specified complete response (CR), CR with incomplete blood count recovery (CRi), nodular partial response (nPR), partial response (PR), or PR with lymphocytosis (PRL) evaluated in accordance with the 2008 IWCLL criteria (Halleck et al). Participants who did not have any postbaseline response assessment were considered as non-responders. This table is based on response assessments performed on or prior to initiation of subsequent antineoplastic therapy or, if applicable, reintroduction of study treatment, whichever occurs earlier. Kaplan-Meier estimate.
  Median follow up duration for the individual MRD Cohort treatment arms: Confirmed uMRD Ibrutinib arm 69.1 months; Confirmed uMRD Placebo arm 67.4 months; uMRD Not Confirmed Ibrutinib arm 47.9 months; uMRD Not Confirmed Ibrutinib + Venetoclax arm 47.9 months.
Time Frame: as for outcome 3
Population: MRD Cohort - All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MRD Cohort: All Treated: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants who completed the planned pre-randomization treatment were eligible to be randomized according to their confirmed undetectable minimal residual disease (uMRD) status: Participants with confirmed uMRD were randomized to receive blinded ibrutinib 420 mg or placebo orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg or open-label ibrutinib 420 mg plus venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. The venetoclax could be administered cumulative from pre-randomization to randomization phase at the dose of 400 mg/day for up to approximately 2 years, or earlier PD or unacceptable toxicity.
- MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded): Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants with confirmed uMRD were randomized to receive ibrutinib 420 mg orally once daily on a continuous schedule until MRD-positive relapse, PD, or unacceptable toxicity, whichever was earlier. After MRD-positive relapse or disease progression (PD) by iwCLL criteria, participants could reintroduce 400 mg venetoclax with a 5-week ramp up. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative), or earlier PD or unacceptable toxicity.
- MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded): Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants with confirmed uMRD were randomized to receive placebo orally once daily on a continuous schedule until MRD-positive relapse, PD or unacceptable toxicity, whichever was earlier. If MRD-positive relapse or PD is confirmed after restaging per iwCLL criteria, participants could first reintroduce oral daily ibrutinib with the option of subsequently reintroducing 400 mg venetoclax with a 5-week ramp up, if subsequent disease relapse per iwCLL criteria occurs after ibrutinib reintroduction. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative), or earlier PD or unacceptable toxicity.
- MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. In case of confirmed PD after restaging per iwCLL criteria, participants could continue ibrutinib and reintroduce venetoclax treatment. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) or earlier PD or unacceptable toxicity.
- MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. In case of confirmed PD after restaging per iwCLL criteria, participants could continue ibrutinib and reintroduce venetoclax treatment. If venetoclax was reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) or earlier PD or unacceptable toxicity.
Arm/Group | MRD Cohort: All Treated | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded) | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 164 | 43 | 43 | 31 | 32
percentage of participants | 97.0 [94.3 to 99.6] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

5. Secondary Outcome: MRD Cohort: Duration of Response (DOR) at 42 Months Landmark Time
Description: Duration of response was calculated for participants achieving a response (CR, CRi, nPR, PR) based on 2008 IWCLL response criteria (Halleck et al.) and defined as the interval between the date of initial documentation of a response including PR with lymphocytosis, until disease progression (PD) or death from any cause, whichever occurred first. As the median DOR was not reached as of 67.0 months study follow-up, the Kaplan-Meier estimate of DOR at 42 months landmark time was presented.
  Median follow up duration for the individual MRD Cohort treatment arms: Confirmed uMRD Ibrutinib arm 69.1 months; Confirmed uMRD Placebo arm 67.4 months; uMRD Not Confirmed Ibrutinib arm 47.9 months; uMRD Not Confirmed Ibrutinib + Venetoclax arm 47.9 months.
Time Frame: From initial documentation of a response until PD or death from any cause, whichever occurs first, for an overall median follow-up of 67.0 months. (Median follow up duration for the individual MRD Cohort treatment arms listed above.)
Population: MRD Cohort: Participants who achieved PR or better
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MRD Cohort: All Treated | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded) | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 159 | 43 | 43 | 31 | 32
percentage of participants | 93.5 [88.2 to 96.4] | 97.6 [84.3 to 99.7] | 93.0 [79.7 to 97.7] | 96.7 [78.6 to 99.5] | 93.2 [75.5 to 98.3]

6. Secondary Outcome: MRD Cohort: MRD-Negativity Rate
Description: MRD negativity rate is defined as the percentage of participants achieving MRD negativity, which is defined as <1 CLL cell per 10,000 leukocytes (<1 x 10^-4) as assessed by flow cytometry of a peripheral blood (PB) or bone marrow (BM) aspirate sample per central laboratory on or prior to initiation of subsequent antineoplastic therapy or, if applicable, reintroduction of study treatment, whichever occurs earlier.
  Median follow up duration for the individual MRD Cohort treatment arms: Confirmed uMRD Ibrutinib arm 69.1 months; Confirmed uMRD Placebo arm 67.4 months; uMRD Not Confirmed Ibrutinib arm 47.9 months; uMRD Not Confirmed Ibrutinib + Venetoclax arm 47.9 months.
Time Frame: From randomization date until before any subsequent antineoplastic therapy, for an overall median follow-up of 67.0 months. (Median follow up duration for the individual MRD Cohort treatment arms listed above.)
Population: MRD All Treated Population; participants with an assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MRD Cohort/uMRD Not Confirmed: All Participants: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg or open-label ibrutinib 420 mg plus venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier.
Arm/Group | MRD Cohort: All Treated | MRD Cohort/uMRD Not Confirmed: All Participants | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 164 | 63 | 31 | 32
percentage of participants
  PB or BM: number analyzed (Participants) | 134 | 41 | 16 | 25
  PB or BM | 81.7 [75.8 to 87.6] | 65.1 [53.3 to 76.9] | 51.6 [34.0 to 69.2] | 78.1 [63.8 to 92.4]
  BM: number analyzed (Participants) | 127 | 35 | 13 | 22
  BM | 77.4 [71.0 to 83.8] | 55.6 [43.3 to 67.8] | 41.9 [24.6 to 59.3] | 68.8 [52.7 to 84.8]
  PB: number analyzed (Participants) | 131 | 38 | 15 | 23
  PB | 79.9 [73.7 to 86.0] | 60.3 [48.2 to 72.4] | 48.4 [30.8 to 66.0] | 71.9 [56.3 to 87.5]

7. Secondary Outcome: MRD Cohort: Tumor Lysis Syndrome (TLS) Risk Reduction Rate With 3-Cycle Ibrutinib Lead-In (Percentage of Participants No Longer High Risk After 3-cycle Lead-in)
Description: TLS risk reduction was summarized by the percentage of participants with TLS risk reduced from high at baseline to medium or low after ibrutinib lead-in. A reduction in TLS risk from high risk to medium or low risk is clinically meaningful because there is a reduction in the extent of TLS monitoring and risk of hospitalization. TLS risk category is defined as the tumor burden category, where: Low=All lymph nodes (LN) < 5 cm AND absolute lymphocyte count (ALC) < 25 x 10^9/L; Medium=Any LN 5 cm to < 10 cm OR ALC ≥ 25 x 10^9/L; High=Any LN ≥ 10 cm OR ALC ≥ 25 x10^9/L AND any LN ≥ 5 cm.
Time Frame: Baseline, and last post-baseline value on or prior to venetoclax first dose date (cycle 4 day 1) or, for participants who never received venetoclax, the post-baseline value closest to cycle 4 day 1 (i.e. 84 days after the first dose date of ibrutinib).
Population: MRD Cohort: All Treated Population with baseline TLS high risk
Measure: Number; unit: percentage of participants
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 40
percentage of participants | 90.0

8. Secondary Outcome: MRD Cohort: Kaplan-Meier Estimate of Progression Free Survival (PFS) Rate at 48 Months Landmark Time
Description: PFS was defined as time from the first dose date of study treatment until disease progression (PD) or death from any cause, whichever occurs first. Assessment of PD was conducted in accordance with the 2008 IWCLL criteria (Halleck et al). As the median PFS was not reached as of the overall median 67.0 months study follow-up, the Kaplan-Meier estimate of PFS rate at 48 months landmark time was presented.
  Median follow up duration for the individual MRD Cohort treatment arms: Confirmed uMRD Ibrutinib arm 69.1 months; Confirmed uMRD Placebo arm 67.4 months; uMRD Not Confirmed Ibrutinib arm 47.9 months; uMRD Not Confirmed Ibrutinib + Venetoclax arm 47.9 months.
Time Frame: From the first dose of ibrutinib to the first confirmed PD or death, for an overall median follow-up of 67.0 months. (Median follow up duration for the individual MRD Cohort treatment arms listed above.)
Population: MRD Cohort - All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib: Participants received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg orally once daily on a continuous schedule until PD or unacceptable toxicity, whichever was earlier. In case of confirmed PD after restaging per iwCLL criteria, participants could continue ibrutinib and reintroduce venetoclax treatment. If venetoclax was to be reintroduced, venetoclax treatment was to continue at the dose of 400 mg/day for up to approximately 2 years (cumulative) or earlier PD or unacceptable toxicity.
Arm/Group | MRD Cohort: All Treated | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded) | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 164 | 43 | 43 | 31 | 32
percentage of participants | 90.9 [85.1 to 94.5] | 97.6 [84.3 to 99.7] | 88.2 [73.9 to 94.9] | 93.3 [75.9 to 98.3] | 93.2 [75.5 to 98.3]

9. Secondary Outcome: MRD Cohort: Kaplan-Meier Estimate of Overall Survival (OS) Rate at 48 Months Landmark Time
Description: OS is defined as the time from the first dose date of study treatment until date of death due to any cause. As the median OS was not reached as of the overall median 67.0 months study follow-up, the Kaplan-Meier estimate of OS rate at 48 months landmark time was presented.
  Median follow up duration for the individual MRD Cohort treatment arms: Confirmed uMRD: Randomized to Ibrutinib=69.1 months; Confirmed uMRD: Randomized to Placebo=67.4 months; uMRD Not Confirmed: Randomized to Open-Label Ibrutinib=47.9 months; uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax=47.9 months.
Time Frame: From the first dose of ibrutinib to time of death, for an overall median follow-up of 67.0 months. (Median follow up duration for the individual MRD Cohort treatment arms listed above.)
Population: MRD Cohort - All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MRD Cohort: All Treated | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded) | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 164 | 43 | 43 | 31 | 32
percentage of participants | 98.0 [94.0 to 99.4] | 97.6 [84.3 to 99.7] | 100.0 [100.0 to 100.0] | 96.7 [78.6 to 99.5] | 100.0 [100.0 to 100.0]

10. Secondary Outcome: MRD Cohort: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs), and Discontinuations Due to TEAEs
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires unplanned in-patient hospitalization >24 hours or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event. Severity of events were graded according to the Common Terminology Criteria for Adverse Events version 4.03: mild=grade1, moderate=grade 2, severe=grade 3, life-threatening=grade 4, death=grade 5. Causal relation of study drug and event was assessed as not related, unlikely, possibly or probably related to the study drug.
Time Frame: From first dose until 30 days following last dose of study drug. Overall median treatment duration for the MRD cohort was 45.1 months.
Population: All Treated Population
Measure: Number; unit: percentage of participants
Arm/Group | MRD Cohort: All Treated | MRD Cohort/Confirmed uMRD: Randomized to Ibrutinib (Blinded) | MRD Cohort/Confirmed uMRD: Randomized to Placebo (Blinded) | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib | MRD Cohort/uMRD Not Confirmed: Randomized to Open-Label Ibrutinib + Venetoclax
Number analyzed (Participants) | 164 | 43 | 43 | 31 | 32
percentage of participants
  Any TEAE | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Any Grade >=3 TEAE | 75.6 | 83.7 | 72.1 | 71.0 | 78.1
  Any Ibrutinib (Ibr)-Related TEAE | 95.7 | 97.7 | 93.0 | 96.8 | 93.8
  Any Grade >=3 Ibrutinib-Related TEAE | 57.9 | 55.8 | 51.2 | 61.3 | 62.5
  Any Venetoclax (Ven)-Related TEAE | 81.1 | 88.4 | 76.7 | 80.6 | 96.9
  Any Grade >=3 Venetoclax-Related TEAE | 44.5 | 51.2 | 34.9 | 45.2 | 56.3
  Any TEAE Leading to Ibr or Ven Discontinuation | 15.9 | 16.3 | 0 | 9.7 | 12.5
  Any TEAE Leading to Ibr or Ven Discontinuation: Ibr Only | 10.4 | 14.0 | 0 | 9.7 | 3.1
  Any TEAE Leading to Ibr or Ven Discontinuation: Ven Only | 1.2 | 2.3 | 0 | 0 | 0
  Any TEAE Leading to Ibr or Ven Discontinuation: Both Ibr and Ven | 4.3 | 0 | 0 | 0 | 9.4
  Any TEAE Leading to Ibr or Ven Dose Reduction | 26.2 | 23.3 | 25.6 | 25.8 | 34.4
  Any TEAE Leading to Ibr Only Dose Reduction | 16.5 | 16.3 | 11.6 | 19.4 | 25.0
  Any TEAE Leading to Ven Only Dose Reduction | 4.9 | 2.3 | 11.6 | 0 | 3.1
  Any TEAE Leading to Both Ibr and Ven Dose Reduction | 4.9 | 4.7 | 2.3 | 6.5 | 6.3
  Any SAE | 34.1 | 34.9 | 32.6 | 41.9 | 37.5
  Any Grade >= 3 SAE | 28.7 | 32.6 | 27.9 | 32.3 | 28.1
  Any SAE Related to Ibr or Ven | 20.1 | 18.6 | 14.0 | 25.8 | 21.9
  Any Ibr-related SAE | 17.1 | 14.0 | 11.6 | 22.6 | 18.8
  Any Ven-related SAE | 6.7 | 4.7 | 7.0 | 12.9 | 6.3
  Fatal TEAE | 1.2 | 2.3 | 0 | 3.2 | 0
  Major Hemorrhage TEAE | 2.4 | 2.3 | 0 | 3.2 | 6.3
  Grade >= 3 Major Hemorrhage TEAE | 1.8 | 2.3 | 0 | 3.2 | 3.1
  Major Hemorrhage SAE | 2.4 | 2.3 | 0 | 3.2 | 6.3

11. Secondary Outcome: FD Cohort: ORR
Description: ORR is defined as the percentage of participants who achieve a best overall response CR, CRi, nPR, PR, or PRL as evaluated by investigator using 2008 IWCLL criteria (Halleck et al.). Participants who did not have any postbaseline response assessment were considered as non-responders. This table is based on response assessments performed on or prior to initiation of subsequent antineoplastic therapy or, if applicable, reintroduction of study treatment, whichever occurs earlier. Kaplan-Meier estimate.
Time Frame: From the first dose of ibrutinib to the first confirmed PD, for a median follow-up of 69.0 months.
Population: FD Cohort: All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FD Cohort, Non-Del 17p Population | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 136 | 159
percentage of participants | 95.6 [92.1 to 99.0] | 96.2 [93.3 to 99.2]

12. Secondary Outcome: FD Cohort: DOR at 60 Months Landmark Time
Description: Duration of response was calculated for participants achieving a response (CR, CRi, nPR, PR) based on 2008 IWCLL response criteria (Halleck et al.) and defined as the interval between the date of initial documentation of a response including PR with lymphocytosis, until disease progression (PD) or death from any cause, whichever occurred first. As the median DOR was not reached as of the median 27.9 months study follow-up, the Kaplan-Meier estimate of DOR at 60 months landmark time was presented.
Time Frame: From initial documentation of a response until PD or death from any cause, whichever occurs first, for a median follow-up of 69.0 months.
Population: FD Cohort: Participants who achieved PR or better.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FD Cohort, Non-Del 17p Population | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 130 | 153
percentage of participants | 63.6 [54.4 to 71.4] | 60.5 [52.0 to 68.0]

13. Secondary Outcome: FD Cohort: MRD Negativity Rate
Description: MRD negativity rate is defined as the percentage of participants achieving MRD negativity, which is defined as <1 CLL cell per 10,000 leukocytes (<1 x 10^-4) as assessed by flow cytometry of a peripheral blood (PB) or bone marrow (BM) aspirate sample per central laboratory on or prior to initiation of subsequent antineoplastic therapy or, if applicable, reintroduction of study treatment, whichever occurs earlier.
Time Frame: From randomization date until before any subsequent antineoplastic therapy, for a median follow-up of 69.0 months.
Population: FD Cohort - All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FD Cohort, Non-Del 17p Population | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 136 | 159
percentage of participants
  BM or PB | 78.7 [71.8 to 85.6] | 78.6 [72.2 to 85.0]
  BM | 61.8 [53.6 to 69.9] | 59.7 [52.1 to 67.4]
  PB | 76.5 [69.3 to 83.6] | 76.7 [70.2 to 83.3]

14. Secondary Outcome: FD Cohort: Kaplan-Meier Estimate of PFS Rate at 66 Months Landmark Time
Description: PFS was defined as time from the first dose date of study treatment until disease progression (PD) or death from any cause, whichever occurs first. Assessment of PD was conducted in accordance with the 2008 IWCLL criteria (Halleck et al). As the median PFS was not reached as of the median 69.0 months study follow-up, the Kaplan-Meier estimate of PFS rate at 66 months landmark time was presented.
Time Frame: From the first dose of ibrutinib to the first confirmed PD or death, for an median follow-up of 69.0 months.
Population: FD Cohort - All Treated Population
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | FD Cohort, Non-Del 17p Population | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 136 | 159
percentage of participants | 63.2 [54.1 to 71.0] | 60.2 [51.7 to 67.7]

15. Secondary Outcome: FD Cohort: Kaplan-Meier Estimate of OS Rate at 66 Months Landmark Time
Description: OS is defined as the time from the first dose date of study treatment until date of death due to any cause. As the median OS was not reached as of the median 69.0 months study follow-up, the Kaplan-Meier estimate of OS rate at 66 months landmark time was presented.
Time Frame: From the first dose of ibrutinib to time of death, for a median follow-up of 69.0 months.
Population: FD Cohort - All Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FD Cohort, Non-Del 17p Population | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 136 | 159
percentage of participants | 96.9 [92.1 to 98.8] | 96.1 [91.4 to 98.2]

16. Secondary Outcome: FD Cohort: TLS Risk Reduction Rate With 3-Cycle Ibrutinib Lead-In (Percentage of Participants No Longer High Risk After 3-cycle Lead-in)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: FD Cohort: All Treated Population with baseline TLS high risk
Measure: Number; unit: percentage of participants
Arm/Group | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 34
percentage of participants | 94.1

17. Secondary Outcome: FD Cohort: Percentage of Participants With TEAEs, Treatment-Emergent SAEs, and Discontinuations Due to TEAEs
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires unplanned in-patient hospitalization >24 hours or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event. Severity of events were graded according to the Common Terminology Criteria for Adverse Events version 4.03: mild=grade1, moderate=grade 2, severe=grade 3, life-threatening=grade 4, death=grade 5. Causal relation of study drug and event was assessed as not related, unlikely, possibly or probably related to the study drug.
Time Frame: From first dose until 30 days following last dose of study drug. Overall median treatment duration for the FD cohort was 13.8 months.
Population: FD Cohort: All Treated Population
Measure: Number; unit: percentage of participants
Arm/Group | Fixed Duration (FD) Cohort: All Treated
Number analyzed (Participants) | 159
percentage of participants
  Any TEAE | 99.4
  Any Grade >=3 TEAE | 62.3
  Any Ibrutinib (Ibr)-Related TEAE | 92.5
  Any Grade >=3 Ibrutinib-Related TEAE | 44.7
  Any Venetoclax (Ven)-Related TEAE | 84.3
  Any Grade >=3 Venetoclax-Related TEAE | 45.3
  Any TEAE Leading to Ibr or Ven Discontinuation | 5.0
  Any TEAE Leading to Ibr or Ven Discontinuation: Ibr Only | 3.1
  Any TEAE Leading to Ibr or Ven Discontinuation: Ven Only | 0
  Any TEAE Leading to Ibr or Ven Discontinuation: Both Ibr and Ven | 1.9
  Any TEAE Leading to Ibr or Ven Dose Reduction | 20.8
  Any TEAE Leading to Ibr Only Dose Reduction | 5.7
  Any TEAE Leading to Ven Only Dose Reduction | 11.3
  Any TEAE Leading to Both Ibr and Ven Dose Reduction | 3.8
  Any SAE | 23.3
  Any Grade >= 3 SAE | 20.1
  Any SAE Related to Ibr or Ven | 13.8
  Any Ibr-related SAE | 11.9
  Any Ven-related SAE | 8.8
  Fatal TEAE | 0.6
  Major Hemorrhage TEAE | 1.9
  Grade >= 3 Major Hemorrhage TEAE | 1.3
  Major Hemorrhage SAE | 1.3

18. Secondary Outcome: MRD Cohort: Pharmacokinetics (PK) of Ibrutinib When Dosed in Combination With Venetoclax: Observed Maximum Concentration (Cmax)
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: MRD Cohort: All treated participants who were evaluable for PK analysis. Data were collected for the MRD cohort only, and without regard to uMRD confirmation status/randomization group, as pre-specified for this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 130
ng/mL | 88.5 (74.3)

19. Secondary Outcome: MRD Cohort: PK of Ibrutinib When Dosed in Combination With Venetoclax: Time to Cmax (Tmax); Time of Last Measurable Concentration (Tlast); Terminal Elimination Half-Life (t1/2,Term)
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: MRD Cohort: All treated participants who were evaluable for each PK analysis. Data were collected for the MRD cohort only, and without regard to uMRD confirmation status/randomization group, as pre-specified for this analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 130
hours
  tmax | 2.00 [0.970 to 7.00]
  tlast | 24.0 [5.75 to 24.0]
  t1/2term | 5.30 [1.47 to 10.5]

20. Secondary Outcome: MRD Cohort: PK of Ibrutinib When Dosed in Combination With Venetoclax: Area Under the Plasma Concentration-Time Curve (AUC) Over the Last 24-hour Dosing Interval (AUC0-24h); AUC From Time Zero to the Time of Last Quantifiable Concentration (AUClast)
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 128
ng*h/mL
  AUC0-24h | 504 (76.3)
  AUClast | 480 (78.5)

21. Secondary Outcome: MRD Cohort: PK of Ibrutinib When Dosed in Combination With Venetoclax: Terminal Elimination Rate Constant (λz)
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 91
1/h | 0.132 (44.5)

22. Secondary Outcome: MRD Cohort: PK of Ibrutinib When Dosed in Combination With Venetoclax: Apparent Total Clearance at Steady-State (CLss/F)
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 128
L/h | 833 (90.9)

23. Secondary Outcome: MRD Cohort: PK of Venetoclax When Dosed in Combination With Ibrutinib: Cmax
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 131
ng/mL | 3034 (56.3)

24. Secondary Outcome: MRD Cohort: PK of Venetoclax When Dosed in Combination With Ibrutinib: Tmax
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 18
Measure: Median (Full Range); unit: hours
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 131
hours | 6.00 [0.00 to 8.08]

25. Secondary Outcome: MRD Cohort: PK of Venetoclax When Dosed in Combination With Ibrutinib: AUC0-24h
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 131
ng*h/mL | 48993 (66.2)

26. Secondary Outcome: MRD Cohort: PK of Venetoclax When Dosed in Combination With Ibrutinib: CLss/F
Time Frame: Cycle 6 Day 1: predose, at dose, 1 h (±15 min), 2 h (±15 min), 4 h (±15 min), 6 h (±15 min), 8 h (±15 min)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | MRD Cohort: All Treated
Number analyzed (Participants) | 131
L/h | 8.16 (69.7)

ADVERSE EVENTS:
Time Frame: From first dose until 30 days following last dose of study drug. Overall median treatment duration was 45.1 months for the MRD cohort and 13.8 months for the FD cohort.
Groups:
- FD Cohort: Pre-Dose: All reported AEs that started prior to the first dose date of any study treatment in the FD Cohort.
- MRD Cohort: Pre-Dose: All reported AEs started prior to the first dose date of any study treatment in the MRD Cohort.
- FD Cohort: All Participants: Participants in the FD Cohort received 420 mg of single agent ibrutinib for first 3 cycles followed by ibrutinib plus venetoclax combination treatment (ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule) for 12 cycles (a cycle is defined by 28 days) or until PD or unacceptable toxicity.
  1. For participants who did not receive any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment over the whole study course.
  2. For participants who received any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment and prior to the first dose date of the reintroduced treatment.
- MRD Cohort: All Participants: Participants in the MRD Cohort received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with confirmed uMRD were randomized to receive blinded ibrutinib 420 mg or placebo orally once daily on a continuous schedule until PD or unacceptable toxicity.
  Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg or open-label ibrutinib 420 mg plus venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity.
  1. For participants who did not receive any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment over the whole study course.
  2. For participants who received any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment and prior to the first dose date of the reintroduced treatment.
- MRD Cohort: Confirmed uMRD (IbrVen->Ibr): Participants in the MRD Cohort with confirmed uMRD received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (prerandomization phase). Participants with confirmed uMRD were randomized to receive ibrutinib 420 mg orally once daily on a continuous schedule until MRD-positive relapse, clinical PD, or unacceptable toxicity.
  1. For participants who did not receive any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment over the whole study course.
  2. For participants who received any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment and prior to the first dose date of the reintroduced treatment.
- MRD Cohort: Confirmed uMRD (IbrVen->Pbo): Participants in the MRD Cohort with confirmed uMRD received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with confirmed uMRD were randomized to receive placebo orally once daily on a continuous schedule until MRD-positive relapse, clinical PD or unacceptable toxicity.
  1. For participants who did not receive any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment over the whole study course.
  2. For participants who received any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment and prior to the first dose date of the reintroduced treatment.
- MRD Cohort: uMRD Not Confirmed (IbrVen->Ibr): Participants in the MRD Cohort with uMRD not confirmed received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg orally once daily on a continuous schedule until PD or unacceptable toxicity.
  1. For participants who did not receive any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment over the whole study course.
  2. For participants who received any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment and prior to the first dose date of the reintroduced treatment.
- MRD Cohort: uMRD Not Confirmed (IbrVen->IbrVen): Participants in the MRD Cohort with uMRD not confirmed received 420 mg of single-agent ibrutinib for the first 3 cycles followed by ibrutinib plus venetoclax combination treatment for at least 12 cycles (a cycle is defined as 28 days) prior to randomization (pre-randomization phase). Participants with uMRD not confirmed were randomized to receive open-label ibrutinib 420 mg and venetoclax 400 mg orally once daily on a continuous schedule until PD or unacceptable toxicity.
  1. For participants who did not receive any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment over the whole study course.
  2. For participants who received any reintroduced treatment, includes all reported AEs started after the first dose date of the first-line treatment and prior to the first dose date of the reintroduced treatment.
- FD Cohort: Reintroduced Ibrutinib: All reported AEs in the FD Cohort that started after the first dose date of reintroduced treatment with ibrutinib.
- FD Cohort: Reintroduced Ibr+Ven: All reported AEs in the FD Cohort that started after the first dose date of reintroduced treatment with ibrutinib + venetoclax.
- MRD Cohort: Reintroduced Ibrutinib: All reported AEs in the MRD Cohort that started after the first dose date of reintroduced treatment with ibrutinib.
- MRD Cohort: Reintroduced Ven + Continued Ibr: All reported AEs in the MRD Cohort that started after the first dose date of reintroduced treatment with venetoclax and continued ibrutinib.
Arm/Group | FD Cohort: Pre-Dose | MRD Cohort: Pre-Dose | FD Cohort: All Participants | MRD Cohort: All Participants | MRD Cohort: Confirmed uMRD (IbrVen->Ibr) | MRD Cohort: Confirmed uMRD (IbrVen->Pbo) | MRD Cohort: uMRD Not Confirmed (IbrVen->Ibr) | MRD Cohort: uMRD Not Confirmed (IbrVen->IbrVen) | FD Cohort: Reintroduced Ibrutinib | FD Cohort: Reintroduced Ibr+Ven | MRD Cohort: Reintroduced Ibrutinib | MRD Cohort: Reintroduced Ven + Continued Ibr
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/164 | 5/159 | 3/164 | 1/43 | 0/43 | 1/31 | 0/32 | 2/18 | 0/11 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/159 | 2/164 | 37/159 | 63/164 | 15/43 | 14/43 | 13/31 | 12/32 | 6/18 | 0/11 | 1/7 | 0/2
Other Adverse Events (participants affected / at risk) | 1/159 | 1/164 | 156/159 | 163/164 | 43/43 | 43/43 | 31/31 | 32/32 | 14/18 | 11/11 | 5/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FD Cohort: Pre-Dose (N=159) | MRD Cohort: Pre-Dose (N=164) | FD Cohort: All Participants (N=159) | MRD Cohort: All Participants (N=164) | MRD Cohort: Confirmed uMRD (IbrVen->Ibr) (N=43) | MRD Cohort: Confirmed uMRD (IbrVen->Pbo) (N=43) | MRD Cohort: uMRD Not Confirmed (IbrVen->Ibr) (N=31) | MRD Cohort: uMRD Not Confirmed (IbrVen->IbrVen) (N=32) | FD Cohort: Reintroduced Ibrutinib (N=18) | FD Cohort: Reintroduced Ibr+Ven (N=11) | MRD Cohort: Reintroduced Ibrutinib (N=7) | MRD Cohort: Reintroduced Ven + Continued Ibr (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 2 (2) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DILATED CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALFORMATION VENOUS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MACULAR OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANTI-NEUTROPHIL CYTOPLASMIC ANTIBODY POSITIVE VASCULITIS (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS ORBITAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER DISSEMINATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PILONIDAL DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 9 (9) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYOMYOSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEST NILE VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA B VIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VESTIBULAR MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ADJUSTMENT DISORDER WITH MIXED ANXIETY AND DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC HAEMATOMA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FD Cohort: Pre-Dose (N=159) | MRD Cohort: Pre-Dose (N=164) | FD Cohort: All Participants (N=159) | MRD Cohort: All Participants (N=164) | MRD Cohort: Confirmed uMRD (IbrVen->Ibr) (N=43) | MRD Cohort: Confirmed uMRD (IbrVen->Pbo) (N=43) | MRD Cohort: uMRD Not Confirmed (IbrVen->Ibr) (N=31) | MRD Cohort: uMRD Not Confirmed (IbrVen->IbrVen) (N=32) | FD Cohort: Reintroduced Ibrutinib (N=18) | FD Cohort: Reintroduced Ibr+Ven (N=11) | MRD Cohort: Reintroduced Ibrutinib (N=7) | MRD Cohort: Reintroduced Ven + Continued Ibr (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 10 (17) | 14 (26) | 5 (10) | 0 (0) | 3 (7) | 5 (7) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 35 (44) | 41 (62) | 12 (19) | 7 (9) | 11 (19) | 8 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 65 (169) | 71 (246) | 24 (107) | 15 (36) | 12 (29) | 14 (54) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 4 (13) | 1 (3) | 0 (0) | 2 (4) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 21 (38) | 33 (72) | 9 (21) | 5 (9) | 5 (12) | 10 (23) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 5 (7) | 13 (18) | 2 (2) | 3 (3) | 3 (3) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 15 (17) | 27 (39) | 11 (18) | 8 (11) | 1 (1) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (6) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (4) | 9 (12) | 2 (2) | 2 (4) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 8 (8) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
RETINAL TEAR (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 13 (15) | 4 (6) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITREOUS HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 10 (12) | 5 (5) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 10 (11) | 15 (21) | 4 (6) | 5 (9) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 13 (16) | 28 (34) | 8 (9) | 10 (11) | 2 (2) | 6 (8) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 14 (15) | 25 (34) | 7 (9) | 5 (6) | 7 (13) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (10) | 7 (10) | 1 (1) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 25 (31) | 34 (47) | 11 (14) | 8 (11) | 9 (12) | 6 (10) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 99 (203) | 119 (435) | 34 (91) | 28 (72) | 23 (56) | 28 (201) | 3 (6) | 4 (7) | 2 (3) | 2 (3)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 8 (8) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 29 (38) | 30 (40) | 10 (11) | 5 (9) | 7 (12) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 9 (9) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 16 (19) | 30 (36) | 10 (11) | 4 (6) | 6 (9) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (8) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLOSSODYNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIP BLISTER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 24 (30) | 19 (31) | 6 (8) | 4 (4) | 6 (10) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 68 (97) | 80 (136) | 21 (40) | 20 (29) | 20 (36) | 12 (22) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALIVARY GLAND ENLARGEMENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 21 (33) | 28 (61) | 9 (13) | 8 (14) | 6 (11) | 3 (20) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 33 (48) | 42 (73) | 13 (26) | 6 (10) | 7 (16) | 11 (14) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 9 (13) | 12 (15) | 2 (2) | 3 (4) | 2 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (8) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 5 (5) | 14 (19) | 4 (5) | 5 (6) | 1 (1) | 4 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 39 (51) | 56 (102) | 14 (25) | 21 (37) | 10 (22) | 7 (12) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 7 (7) | 11 (12) | 4 (5) | 1 (1) | 4 (4) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
INJECTION SITE BRUISING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 7 (7) | 6 (7) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 11 (12) | 22 (34) | 8 (11) | 6 (11) | 3 (4) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 4 (7) | 9 (10) | 0 (0) | 2 (2) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 11 (11) | 6 (6) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 22 (35) | 31 (44) | 10 (12) | 4 (7) | 3 (5) | 10 (13) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 7 (7) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 7 (7) | 14 (19) | 3 (3) | 7 (7) | 0 (0) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 8 (9) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 8 (9) | 29 (38) | 14 (18) | 13 (18) | 2 (2) | 0 (0) | 3 (4) | 2 (2) | 3 (4) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 4 (7) | 0 (0) | 1 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 7 (13) | 4 (10) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 8 (8) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 8 (9) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 10 (10) | 13 (16) | 7 (10) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 7 (8) | 8 (11) | 4 (5) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 6 (7) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 12 (16) | 26 (33) | 7 (11) | 6 (7) | 8 (9) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NOROVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ONYCHOMYCOSIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 7 (8) | 8 (10) | 3 (5) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 14 (23) | 5 (10) | 2 (2) | 3 (3) | 4 (8) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROSTATIC ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 8 (14) | 1 (5) | 6 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SIALOADENITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 10 (17) | 23 (38) | 7 (11) | 4 (7) | 7 (11) | 4 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 6 (7) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 39 (50) | 73 (138) | 21 (44) | 22 (48) | 14 (24) | 11 (15) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 12 (17) | 23 (40) | 8 (15) | 6 (11) | 6 (8) | 3 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 6 (8) | 1 (1) | 1 (1) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 24 (25) | 40 (63) | 10 (14) | 12 (20) | 10 (14) | 6 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 10 (11) | 5 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (5) | 9 (10) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 9 (9) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 6 (6) | 17 (33) | 4 (7) | 5 (6) | 4 (11) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 9 (16) | 17 (24) | 5 (5) | 5 (6) | 4 (7) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 6 (15) | 7 (20) | 1 (1) | 0 (0) | 5 (17) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 7 (8) | 16 (20) | 5 (6) | 4 (4) | 3 (5) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 16 (38) | 5 (6) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 8 (14) | 9 (12) | 5 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 6 (6) | 8 (8) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 7 (18) | 4 (6) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (9) | 19 (23) | 6 (7) | 8 (8) | 4 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (8) | 0 (0) | 0 (0) | 1 (4) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (7) | 9 (12) | 2 (3) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 12 (15) | 3 (6) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (9) | 8 (11) | 4 (4) | 3 (4) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 12 (21) | 15 (25) | 7 (11) | 2 (2) | 1 (2) | 4 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (8) | 11 (20) | 3 (8) | 3 (5) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (15) | 3 (5) | 1 (1) | 1 (2) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (12) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (8) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6) | 8 (9) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 52 (84) | 82 (162) | 23 (48) | 20 (40) | 17 (28) | 16 (34) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 20 (22) | 42 (57) | 11 (12) | 9 (14) | 10 (17) | 9 (11) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 9 (12) | 5 (8) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 47 (66) | 43 (61) | 13 (20) | 11 (17) | 10 (11) | 7 (11) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 23 (30) | 31 (46) | 9 (18) | 9 (11) | 7 (8) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (7) | 12 (12) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 21 (25) | 31 (39) | 5 (5) | 9 (12) | 8 (8) | 8 (13) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (4) | 12 (18) | 4 (6) | 5 (5) | 1 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRAIN FOG (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 27 (34) | 32 (45) | 10 (14) | 9 (11) | 5 (9) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 39 (55) | 52 (92) | 15 (27) | 18 (32) | 8 (16) | 9 (14) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 12 (15) | 3 (3) | 4 (5) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 14 (18) | 4 (4) | 4 (6) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 13 (14) | 4 (4) | 2 (3) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 4 (4) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (6) | 21 (22) | 3 (3) | 6 (7) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 9 (9) | 12 (14) | 3 (3) | 2 (2) | 3 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR SWELLING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 28 (34) | 46 (63) | 15 (20) | 17 (25) | 8 (10) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 11 (11) | 22 (25) | 11 (12) | 6 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 19 (27) | 30 (51) | 10 (18) | 8 (17) | 5 (8) | 6 (7) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 18 (21) | 7 (8) | 4 (5) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 17 (19) | 39 (63) | 10 (16) | 9 (15) | 9 (16) | 10 (14) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 6 (6) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 10 (10) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (7) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 9 (9) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 7 (7) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 5 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 16 (18) | 25 (28) | 10 (13) | 7 (7) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 12 (16) | 7 (10) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (8) | 13 (18) | 2 (2) | 4 (6) | 2 (4) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (6) | 7 (8) | 0 (0) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 15 (18) | 4 (5) | 3 (3) | 5 (6) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 14 (14) | 22 (23) | 5 (5) | 5 (6) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 17 (23) | 25 (35) | 5 (6) | 3 (6) | 6 (9) | 8 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 17 (19) | 21 (30) | 7 (9) | 2 (3) | 3 (4) | 8 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (12) | 19 (23) | 5 (5) | 4 (5) | 3 (5) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 9 (11) | 13 (16) | 3 (5) | 4 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 27 (32) | 29 (38) | 9 (12) | 10 (11) | 5 (9) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 9 (9) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN FRAGILITY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (8) | 13 (16) | 4 (7) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN MASS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 24 (33) | 45 (68) | 15 (26) | 11 (16) | 9 (13) | 8 (10) | 2 (5) | 5 (7) | 3 (4) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT02910583/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT02910583/SAP_001.pdf